CLINICAL TRIAL: NCT06982612
Title: Glycemic Control Following Occupational Work in a Hot Environment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Stephen Mears, Dr - Senior lecturer, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LEON21544
Record Dates: First submitted 2025-05-01; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Plasma Glucose Following Prolonged Heat Exposure
Keywords: heat; plasma glucose; worker; glycemia; OGTT

STUDY DESIGN:
Intervention Model Description: Randomised, crossover design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot condition (Experimental): Light exercise in a hot environment with ad libitum water intake
  Interventions: Other: Hot environment
- Temperate condition (Experimental): Light exercise in a temperate environment with ad libitum water intake
  Interventions: Other: Temperate condition

INTERVENTIONS:
Other: Hot environment — Participants exercising in a 36 degrees celsius environment
  Arms: Hot condition
Other: Temperate condition — Participants exercising in a 18 degrees celsius environment
  Arms: Temperate condition

SUMMARY:
Occupational workers regularly perform physically demanding tasks in hot environments, exposing them to heat stress and potential dehydration. While the physiological impacts of heat exposure are well-documented, its effects on glycemic control remain less understood. Given the rising global temperatures due to climate change and the increasing prevalence of metabolic disorders such as obesity and type 2 diabetes, it is essential to investigate how heat exposure during work influences glycemic regulation. Understanding these interactions will help inform future occupational health guidelines and metabolic health recommendations in physically demanding industries.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Generally fit and healthy
* Participate in endurance or intermittent exercise at least 3 times a week or minimum of 150 minutes moderate intensity activity per week

Exclusion Criteria:

* Under 18 or 45 and over,
* any morbidity or medication that might influence carbohydrate/fat metabolism (i.e., liver/renal/cardiovascular disease) or cycling ability (musculoskeletal injury etc),
* coagulation or bleeding disorders,
* blood-borne illness,
* heart conditions,
* congenital heart disease,
* uncontrolled exercise-induced asthma,
* smoking (including vaping),
* allergies to the products used in the study,
* dieting or restrained eating behaviours.
* Females with amenorrhea would be an exclusion criteria.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose | 8hours
  Measured using colorimetric assay from venous blood samples

SECONDARY OUTCOMES:
Plasma insulin | 8hours
  Measured using ELISA from venous blood samples
Plasma osmolality | 8hours
  Measured using freezing point depression from venous blood samples
Plasma volume change | 8hours
  Determined from haemoglobin and haematocrit measures in blood samples
Urine volume | 8hours
  Determined from urine samples collected before and after exercise
Body mass | 8hours
  Determined from weighing participants before and after exercise
Urine specific gravity/osmolality | 8hours
  Determined from urine samples collected before and after exercise
Rectal temperature | 8hours
  Measured via rectal probe
Blood pressure | 8hours
  Measured via and automated sphygmomanometer
Respiratory gas exchanges | 8hours
  Measured via Douglas bag, gas content and volume
Rate of perceived exertion | 8hours
  using Borg scales (from 6 [no effort] to 20 [maximal effort])
Rate of thermal sensation | 8hours
  using -10 [cold] to +10 [hot] scale.
Feelings of thirst, urge to urinate, GI comfort, and stomach bloatedness | 8hours
  using scales (0 = no feeling, 10 = extreme feeling)

OTHER OUTCOMES:
N-back task for working memory (cognitive function) | 8hours
  The task will comprise three progressively harder memory loads (1-Back, 2-Back, 3-Back). Each stimulus type will be used in all memory loads. Participants will have to respond using the space bar when they see a stimulus that is presented one, two, or three steps previously, dependent on the load condition.
Go/no-go task for response inhibition (cognitive function) | 8hours
  Participants will be instructed to press the space bar when a green image appears onscreen ("go" stimulus) and to inhibit responding when a red image is presented (the "no-go" stimulus). Increased commission error responses (i.e. responding incorrectly on a no-go trial) will indicate reduced response inhibition. Commission errors and correct responses will be measured as indices of performance.
Stroop test | 8hours
  The Stroop Test is a psychological assessment that measures a person's ability to inhibit cognitive interference and control attention. Typically, it involves naming the color of the ink in which a word is printed, even when the word itself names a different color (e.g., the word "red" printed in blue ink). The delay in response time when the word and ink color do not match-known as the Stroop effect-reflects the difficulty of suppressing automatic cognitive processes.

IPD SHARING:
Plan to Share IPD: No